CLINICAL TRIAL: NCT04881890
Title: A Mixed Methods Pilot Study of a Low-Carbohydrate Diabetes Prevention Program Among Veterans With Prediabetes
Brief Title: Low-Carbohydrate Diabetes Prevention Program Among Veterans With Prediabetes
Acronym: VA LC-DPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LIP 20-122
Record Dates: First submitted 2020-11-17; First posted 2021-05-11 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Carbohydrate Diabetes Prevention Program (Experimental): At least 20 individuals with prediabetes will participate in a year-long , group-based program.
  Interventions: Behavioral: Low-Carbohydrate Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diabetes Prevention Program — LC-DPP participants will be instructed to follow ad-libitum very low-carbohydrate, ketogenic diet, which restricts carbohydrate intake (not including fiber) to 20-35 grams per day with the goal of achieving nutritional ketosis. Participants will be encouraged to eat a normal amount of protein (roughly 80-120 grams per day) and to derive the remaining calories from fat. Allowable foods include: meats, fish, poultry, eggs, cheese, seeds, nuts, leafy greens, non-starchy vegetables, and some fruits

SUMMARY:
The investigators will conduct a single-arm mixed methods pilot study to examine the feasibility and acceptability of a low-carbohydrate diabetes prevention program (LC-DPP). The investigators will estimate weight loss as well as the percentage of participants who achieve 5% body weight loss at 6 month and 12 month timepoints. Weight loss from the pilot VA LC-DPP cohort will be compared to weight loss outcomes from previously published DPP studies and the VA MOVE! program. The investigators will also evaluate secondary outcomes including change in physical activity, mental health, psychosocial functioning, and hemoglobin A1c over the 12-month study period. The investigators will also conduct qualitative interviews with participants at 6 and 12 months.

DETAILED DESCRIPTION:
The Veteran population faces high rates of T2DM with estimates surpassing 20% compared to 14% among the general population. Furthermore, an estimated 25% of overweight or obese Veterans have prediabetes and many will progress to T2DM over time. Fortunately, T2DM can be prevented or delayed through dietary and physical activity changes that promote weight loss of ≥5% body weight. To help Veterans lose weight and avoid obesity-related chronic conditions such as T2DM, the VA Health System offers a lifestyle change program, VA MOVE!. Although MOVE! is widely adopted across the VA Health System, weight loss outcomes are modest (range of 0.13-3.3 kg loss over one year) and less than 20% of participants achieve ≥5% weight loss.

Novel strategies are needed to help more Veterans to lose weight and prevent and manage obesity-related conditions. One promising approach may be through a low-carbohydrate dietary intervention. Consistent with historic United States Dietary Guidelines, diabetes prevention clinical trials and their translational group-based programs, including VA MOVE!, recommend a low-fat, calorie-restricted diet. However, the scientific merit of this recommendation has been criticized. Growing evidence supports the efficacy of low-carbohydrate diets (defined <26% total energy from carbohydrate per day) and VLCDs (defined as <10% of total energy from carbohydrate per day) for short-term weight loss, long-term weight maintenance, and improved glycemic control, particularly among individuals with T2DM and insulin resistance.

The objectives of this single-arm mixed methods pilot study are (1) to test the feasibility and acceptability of a low-carbohydrate Diabetes Prevention Program (LC-DPP) among Veterans with prediabetes and (2) to estimate weight loss among LC-DPP participants.

The investigators will recruit approximately 22 patients with body mass index ≥ 25 kg/m2 and prediabetes (defined as hemoglobin A1c [A1c] 5.7-6.4%). Participants will be identified by chart review and invited to participate by postal letter. Individuals that do not opt-out of study contact will be screened for eligibility by telephone call. Interested and eligible participants will be invited to attend an in-person information session. During this session, they will receive information about the dietary intervention; written informed consent will be obtained at this time. Study participants will attend a total of 24 group-based classes over the course of 1-year. Body weight will be measured at each session. At 0, 6, and 12-months, the investigators will measure hemoglobin A1c (HbA1c) and cholesterol levels as well as self-reported measures of quality of life, mood, hunger, cravings, and physical symptoms. Primary outcomes will be feasibility (e.g., enrollment, retention) and acceptability (e.g., session attendance, qualitative feedback). Secondary outcomes will change in weight, achievement of ≥5% body weight loss, change in HbA1c, and change in cholesterol levels. During semi-structured interviewed conducted at 6-months and 12-months, the investigators will explore participants' experiences with the program, barriers to and facilitators of adherence to a low-carbohydrate diet, and perspectives on ways to improve the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight, defined as BMI≥25 kg/m2 [31]
2. HbA1c between 5.7-6.4% drawn within 1 year of the study start date
3. Willingness to participate in group-based classes
4. Able to engage in at least light physical activities such as walking.

Exclusion Criteria:

1. History of type 1 diabetes or type 2 diabetes
2. Current participation in another lifestyle or behavior change program or research study
3. Vegetarian or vegan lifestyle
4. History of bariatric surgery
5. Inability to read, write, or speak English
6. Inability to provide informed consent
7. Women who are pregnant or intend to become pregnant during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Assess recruitment feasibility and interest in the study | Baseline
  This will be calculated by dividing by number of enrolled participants by the number of individuals invited to participate.
Retention of participants in the study | 6 months
  Retention of participants in the study will be determined by the participant completion of surveys
Retention of participants in the study | 12 months
  Retention of participants in the study will be determined by the participant completion of surveys
Session attendance | 6 months
  Attendance will determined by the mean number meetings attended by each participant
Session attendance | 12 months
  Attendance will determined by the mean number meetings attended by each participant
Acceptability of the program by participants | 6 month
  Determined by semi-structured interview responses
Acceptability of the program by participants | 12 month
  Determined by semi-structured interview responses
Adherence with self-weighing | 6 months
  Calculated by dividing the number of self-reported weights by the number of sessions.
Adherence with self-weighing | 12 months
  Calculated by dividing the number of self-reported weights by the number of sessions.
Adherence with physical activity goals | 6 months
  Defined by participants that report at least 150 minutes of physical activity in a week.
Adherence with physical activity goals | 12 months
  Defined by participants that report at least 150 minutes of physical activity in a week.
Adherence with food tracking | 6 months
  Defined by participants that report maintaining a food log.
Adherence with food tracking | 12 months
  Defined by participants that report maintaining a food log.

SECONDARY OUTCOMES:
Change in physical activity measured using the International Physical Activity Questionnaire | 6 months to baseline
  Participants will complete this validated survey. Minimum value: 0, Maximum Value: 9.
Change in physical activity measured using the International Physical Activity Questionnaire | 12 months to baseline
  Participants will complete this validated survey. Minimum value: 0, Maximum Value: 9.
Change in food cravings measured using the Control of Eating Questionnaire | 6 months to baseline
  Participants will complete this validated survey. Minimum value: 0, Maximum Value: 100.
Change in food cravings measured using the Control of Eating Questionnaire | 12 months to baseline
  Participants will complete this validated survey. Minimum value: 0, Maximum Value: 100.
Change in stress eating measured using the Palatable Eating Motives Scale | 6 months to baseline
  Participants will complete this validated survey.
Change in stress eating measured using the Palatable Eating Motives Scale | 12 months to baseline
  Participants will complete this validated survey
Change in self-reported health measured using the Global Health PROMIS Questionnaire | 6 months to baseline
  Participants will complete this validated survey. Minimum Value: 1. Maximum Value: 5. The higher value indicated a more positive response.
Change in self-reported health measured using the Global Health PROMIS Questionnaire | 12 months to baseline
  Participants will complete this validated survey. Minimum Value: 1. Maximum Value: 5. The higher value indicated a more positive response.
Change in autonomous motivation measured using the Treatment Self-Regulation Questionnaire | 6 months to baseline
  Participants will complete this validated survey. Minimum Value: 1. Maximum Value: 7. The higher value indicated a more positive response.
Change in autonomous motivation measured using the Treatment Self-Regulation Questionnaire | 12 months to baseline
  Participants will complete this validated survey. Minimum Value: 1. Maximum Value: 7. The higher value indicated a more positive response.
Measured change in hemoglobin A1c | 6 months to baseline
  Measured using a laboratory blood draw
Measured change in hemoglobin A1c | 12 months to baseline
  Measured using a laboratory blood draw
Change in hemoglobin A1c | 6 months to baseline
  Baseline A1c will be subtracted from the 6 month A1c.
Change in hemoglobin A1c | 12 months to baseline
  Baseline A1c will be subtracted from the 12 month A1c.
Change in lipid levels | 6 months to baseline
  Baseline lipid levels will be subtracted from the 6 month lipid level.
Change in lipid levels | 12 months to baseline
  Baseline lipid levels will be subtracted from the 12 month lipid level.
Percentage of participants who achieve weight loss goal | 6 month
  Determined by the number of participants who lose at least 5% of their body weight during the study
Percentage of participants who achieve weight loss goal | 12 month
  Determined by the number of participants who lose at least 5% of their body weight during the study
Change in body weight per participant over the study period | 6 months to baseline
  Determined by subtracting the patients baseline weight from their weight at 6 months.
Change in body weight per participant over the study period | 12 months to baseline
  Determined by subtracting the patients baseline weight from their weight at 12 months.

OTHER OUTCOMES:
Change in physical symptoms | 6 months to baseline
  Participants will respond to exploratory survey questions about physical symptoms created by the study team.
Change in physical symptoms | 12 months to baseline
  Participants will respond to exploratory survey questions about physical symptoms created by the study team.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veteran Affairs, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griauzde DH, Hershey C, Michaels J, Evans RR, Richardson CR, Heisler M, Kullgren JT, Saslow LR. A very low-carbohydrate diabetes prevention program for veterans with prediabetes: a single-arm mixed methods pilot study. Front Nutr. 2023 May 17;10:1069266. doi: 10.3389/fnut.2023.1069266. eCollection 2023. PMID 37266128

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04881890/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04881890/SAP_001.pdf